CLINICAL TRIAL: NCT04299477
Title: EVALUATION OF THE EFFETCS OF NON-SURGICAL PERIODONTAL TREATMENT ON SALIVARY BIOMARKERS OF PATIENTS UNDERGOING BISPHOSPHONATE THERAPY
Brief Title: THE EFFETCS OF NON-SURGICAL PERIODONTAL TREATMENT ON SALIVARY BIOMARKERS OF PATIENTS WITH OSTEOPOROSIS AND PERIODONTITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Basak Karasu, Principal Investigator, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/26120
Record Dates: First submitted 2020-01-22; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis; Periodontitis
Keywords: non-surgical periodontal treatment; bisphosphonates; interleukin-1β; interleukin-17; 8-hydroxydeoxyguanosine; alkaline phosphatase
MeSH Terms: conditions — Osteoporosis; Periodontitis

STUDY DESIGN:
Intervention Model Description: 25 patients with periodontitis (P) and osteoporosis (group 1), 25 systemically healthy patients with P (group 2) and 25 systemically and periodontally healthy individuals (group 3) were enrolled in this study.
  Individuals were periodontally examined at baseline, 1 month and 3 months following the non-surgical periodontal therapy.
  Participants in group 1 and 2 received non-surgical periodontal therapy including supra- and subgingival scaling, and root planning.Patients were advised and instructed to perform oral care twice a day, use interdental toothbrushes once a day regularly. No scaling and root planning was performed in the group 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with periodontitis and osteoporosis (Experimental): Group 1 : Patients who have periodontitis and osteoporosis prescribed with bisphosphonates
  Interventions: Procedure: non-surgical periodontal treatment
- Systemically healthy patients with periodontitis (Experimental): Group 2: Patients who have no systemic diseases but diagnosed as periodontitis
  Interventions: Procedure: non-surgical periodontal treatment
- Systemically and periodontally healthy individuals (No Intervention): Group 3: Healthy controls

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — supra- and subgingival scaling, and root planning
  Arms: Patients with periodontitis and osteoporosis; Systemically healthy patients with periodontitis

SUMMARY:
Inflammatory mediators in periodontitis may lead to elevated systemic cytokine levels, resulting in increased bone resorption including the jaws. Osteoporosis may have an influence on the periodontal condition of post-menopausal women and the risk for periodontal disease may increase due to osteoporosis. The hypothesis of the study was that non-surgical periodontal treatment and medical treatment of osteoporosis by bisphosphonates may improve the clinical outcomes and decrease salivary levels of IL-1β, IL-17, ALP and 8-OHdG. Therefore, the aim of this study was to evaluate the mechanism of bi-directional relationship between osteoporosis and periodontal diseases and to investigate the outcomes of non-surgical periodontal treatment with regard to salivary levels of IL-1β, IL-17, 8-OHdG and ALP in patients with periodontitis and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* The participants were postmenopausal patients defined as absence of menstruation for at least 12 months.
* Patients with periodontitis;
* Patients who had no systemic diseases and were periodontally healthy (no attachment loss),
* Patients who were treated with oral bisphosphonate at least one year (70 mg tablet once weekly)

Exclusion Criteria:

* if they had received any periodontal treatment in the preceding three months,
* if they were pregnant or in the period of lactation,
* if they had systemic diseases that may interfere with normal healing mechanism,
* if they had taken antibiotics, anticonvulsants, immunosuppressants, calcium channel blockers in the preceding six months.
* Smokers

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
salivary levels of IL-1β at baseline | baseline
  evaluation of the salivary levels of IL-1β in g/ml
salivary levels of IL-1β at 1-month | 1-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of IL-1β in g/ml
salivary levels of IL-1β at 3-month | 3-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of IL-1β in g/ml
salivary levels of IL-17 baseline | baseline
  evaluation of the salivary levels of IL-17 in g/ml
salivary levels of IL-17 at 1-month | 1-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of IL-17 in g/ml
salivary levels of IL-17 at 3-month | 3-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of IL-17 in g/ml
salivary levels of alkaline phosphatase at baseline | baseline
  evaluation of the salivary levels of alkaline phosphatase in g/ml
salivary levels of alkaline phosphatase at 1-month | 1-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of alkaline phosphatase in g/ml
salivary levels of alkaline phosphatase at 3-month | 3-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of alkaline phosphatase in g/ml
salivary levels of 8-hydroxydeoxyguanosine at baseline | baseline
  evaluation of the salivary levels of 8-hydroxydeoxyguanosine in g/ml
salivary levels of 8-hydroxydeoxyguanosine at 1-month | 1-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of 8-hydroxydeoxyguanosine in g/ml
salivary levels of 8-hydroxydeoxyguanosine at 3-month | 3-month follow-up after non-surgical periodontal therapy
  evaluation of the salivary levels of 8-hydroxydeoxyguanosine in g/ml

SECONDARY OUTCOMES:
Plaque index | baseline, 1- and 3-month follow- up.
  Plaque index scores assessed at baseline and at 1 month and 3 months after non-surgical periodontal therapy
gingival index | baseline, 1- and 3-month follow- up.
  gingival index scores assessed at baseline and at 1 month and 3 months after non-surgical periodontal therapy
bleeding on probing | baseline, 1- and 3-month follow- up.
  bleeding on probing scores assessed at baseline and at 1 month and 3 months after non-surgical periodontal therapy
probing depth | baseline, 1- and 3-month follow- up.
  probing depth scores assessed at baseline and at 1 month and 3 months after non-surgical periodontal therapy
clinical attachment level | baseline, 1- and 3-month follow- up.
  clinical attachment level scores assessed at baseline and at 1 month and 3 months after non-surgical periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Basak Karasu, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Cankaya, Turkey (Türkiye)